CLINICAL TRIAL: NCT02621775
Title: Effectiveness of Two Stress Management Programs in the Adaptation Disorder With Anxiety (ADA) : Computer-based or Face- to -Face to Face Versus Control Group.Open Multicenter Prospective Randomized Controlled Therapeutic 3 Parallel Groups
Brief Title: Effectiveness of Two Stress Management Programs in Adaptation Disorder With Anxiety (ADA)
Acronym: Seren@ctif
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014_36; 2015-A00098-41 (Other: ID-RCB number, ANSM); PHRCI_2014 (Other: PHRC number, DGOS)
Record Dates: First submitted 2015-11-26; First posted 2015-12-03 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2019-06

CONDITIONS: Adjustment Disorders; Psychological Stress
Keywords: Stress management; Cognitive behavioural therapy (CBT); Self-help; e-health; Adjustment disorder with anxiety
MeSH Terms: conditions — Adjustment Disorders; Stress, Psychological | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Computer-based stress management program (Experimental): Immediate e-learning condition with minimal contact (n =40),
  Interventions: Behavioral: Computer-based stress management program
- Stress management in face-to-face (Experimental): Immediate treatment in face - to- face (n = 40)
  Interventions: Behavioral: Stress management in face-to-face
- Waiting list (Other): Waiting list (n=40)
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Computer-based stress management program — The program includes 5 one hour weekly sessions that patient follow from a web site accessible from a computer in our unit. He benefits from a minimal contact with a medical member of staff before and after every session. The duration of each session is about one hour. To avoid internet connexion problem between session it is supplied to the patient, from the first session an USB key (Universal Serial Bus) containing videos, audio files, self help book, portfolio in the form of e-guide, log book with the program of the exercises to be realized between two session of the five sessions program. The patient is encouraged to practice a twenty-minutes daily exercises five or six days per week.
  Other Names: Seren@ctif
  Arms: Computer-based stress management program
Behavioral: Stress management in face-to-face — The program includes 5 forty-five minutes weekly session with a therapist (psychologist graduate of a master of cognitive and emotional therapy with a minimal of one year of practice in CBT and CBSM (Cognitive-Behavioral Stress Management ). Information, exercises and homework assignments are delivered by the therapist without self help support.
  Arms: Stress management in face-to-face
Other: Waiting list — The patients are followed by their General Practitioners without change in treatment .
  Arms: Waiting list

SUMMARY:
The aim of this study was to assess the effects of a 5-week standardized cognitive behavioral treatment of stress management conducted via e-learning or face-to-face on patients responding to the diagnosis of adjustment disorder with anxiety (ADA) according to the DSM- 5 (Diagnostic and Statistical Manual of Mental Disorders Fifth Edition) criteria .

DETAILED DESCRIPTION:
The program includes 5 weekly sessions that the patient follows. It is based on standard CBT (Cognitive Behavioural Therapy) principles and includes five modules (information about stress and stress reaction and assessment; deep respiration and relaxation techniques; cognitive re-structuration; mindfulness and acceptation; behavioral skills as solving problem, time management, healthy behaviors, problem solving and emotion regulation …).

* In internet-based group patient benefits from a minimal contact with a medical member of staff before and after every session. It is supplied to the patient, from the first session an USB key containing videos, audio files, help-self book portfolio in the form of e-guide, log books with the program of the exercises to be realized between two session of the 5 sessions program. The patient is encouraged to practice a twenty-minutes daily of exercises five or six days per week.
* In face-to-face group, patient receive the same program with a therapist in 5 weekly sessions without digital supports.

ELIGIBILITY:
Inclusion Criteria:

* Adjustment disorder with anxiety (ADA) according DSM-5 (The diagnosis was made according to the MINI questionnaire).
* Subscore anxiety > 10, subscore depression < 10 at Hospital Anxiety Depression Scale (HADS)
* Computer at home

Exclusion Criteria:

* Subscore anxiety < 10, subscore depression > 10 at Hospital Anxiety Depression Scale (HADS)
* No others current psychiatric diagnostic according DSM- 5
* No suicidal ideation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Score of State-Trait Anxiety Inventory (STAI-S), | Between baseline and 2 month of use
  self-administered questionnaire of 20 items side on 4 levels from 'not at all' to one side "many" side 4 (total score of 20-80). It measures an intensity of more anxiety and is not related to an anxiety disorder.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale (HAD), | at 2 months, at 6 months
  The scale allows to detect anxiety and depression using 14 items rated from 0-3.
The Penn-State Worry Questionnaire (PSWQ), | at 2 months, at 6 months
  Self-Assessment Questionnaire consisting of 16 items, measuring the general tendency to worry.
The Perceived Stress Scale (PSS) | at 2 months, at 6 months
  Two dimensions emerge from this scale: the overflow and perceived self-efficacy.
Visual Analogue Scale for stress (VAS-stress) | at 2 months, at 6 months
The Beck depression inventory (BDI-21) | at 2 months, at 6 months
  Self-assessment questionnaire measuring the severity of depression

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Servant, MD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Centre Pinel, Amiens
  - Centre Esquirol CHU de Caen, Caen
  - CHRU , Hôpital FONTAN, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Day V, McGrath PJ, Wojtowicz M. Internet-based guided self-help for university students with anxiety, depression and stress: a randomized controlled clinical trial. Behav Res Ther. 2013 Jul;51(7):344-51. doi: 10.1016/j.brat.2013.03.003. Epub 2013 Mar 28. PMID 23639300
- [Background] Drozd F, Raeder S, Kraft P, Bjorkli CA. Multilevel growth curve analyses of treatment effects of a Web-based intervention for stress reduction: randomized controlled trial. J Med Internet Res. 2013 Apr 22;15(4):e84. doi: 10.2196/jmir.2570. PMID 23607962
- [Background] Eisen KP, Allen GJ, Bollash M, Pescatello LS. Stress management in the workplace: A comparison of a computer-based and an in-person stress-management intervention. Comput Hum Behav. 2008 Mar;24(2):486-96.
- [Background] Grime PR. Computerized cognitive behavioural therapy at work: a randomized controlled trial in employees with recent stress-related absenteeism. Occup Med (Lond). 2004 Aug;54(5):353-9. doi: 10.1093/occmed/kqh077. PMID 15289593
- [Background] Rose RD, Buckey JC Jr, Zbozinek TD, Motivala SJ, Glenn DE, Cartreine JA, Craske MG. A randomized controlled trial of a self-guided, multimedia, stress management and resilience training program. Behav Res Ther. 2013 Feb;51(2):106-12. doi: 10.1016/j.brat.2012.11.003. Epub 2012 Nov 21. PMID 23262118
- [Background] Ruwaard J, Lange A, Bouwman M, Broeksteeg J, Schrieken B. E-mailed standardized cognitive behavioural treatment of work-related stress: a randomized controlled trial. Cogn Behav Ther. 2007;36(3):179-92. doi: 10.1080/16506070701381863. PMID 17852171
- [Background] Servant D, Rougegrez L, Barasino O, Demarty AL, Duhamel A, Vaiva G. [Interest of computer-based cognitive behavioral stress management. Feasability of the Seren@ctif program]. Encephale. 2016 Oct;42(5):415-420. doi: 10.1016/j.encep.2016.03.010. Epub 2016 Apr 25. French. PMID 27126141
- [Result] Leterme AC, Behal H, Demarty AL, Barasino O, Rougegrez L, Labreuche J, Duhamel A, Vaiva G, Servant D. A blended cognitive behavioral intervention for patients with adjustment disorder with anxiety: A randomized controlled trial. Internet Interv. 2020 May 25;21:100329. doi: 10.1016/j.invent.2020.100329. eCollection 2020 Sep. PMID 32523873
- [Derived] Servant D, Leterme AC, Barasino O, Rougegrez L, Duhamel A, Vaiva G. Efficacy of Seren@ctif, a Computer-Based Stress Management Program for Patients With Adjustment Disorder With Anxiety: Protocol for a Controlled Trial. JMIR Res Protoc. 2017 Oct 2;6(10):e190. doi: 10.2196/resprot.7976. PMID 28970192